CLINICAL TRIAL: NCT05883709
Title: A Real-world Study Evaluating the Safety and Efficacy of Tafasitamab in Combination With Lenalidomide in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: A Real-world Study of Tafasitamab in Combination With Lenalidomide in Patients withR/R DLBCL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhao Weili (Other)
Responsible Party: Sponsor-Investigator, Zhao Weili, Prof., Ruijin Hospital
Organization: Ruijin Hospital (Other)
Other Study IDs: KY2023-006
Record Dates: First submitted 2023-05-20; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tafasitamab; Lenalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Tafa combination therapy group, which could include Tafa combined with lenalidomide, Tafa combined with Lenalidomide plus BTK inhibitors, Tafa combined with Lenalidomide plus chemotherapy (including ADC)
  Interventions: Drug: Tafasitamab Injection
- Cohort 2: Tafa combination therapy group followed by sequential CAR T or transplantation
  Interventions: Drug: Tafasitamab Injection

INTERVENTIONS:
Drug: Tafasitamab Injection — The combination of Tafasitamab and lenalidomide based treatment was selected according to the specific conditions of patients
  Other Names: lenalidomide

SUMMARY:
To evaluate the real-world efficacy of Tafasitamab combined with Lenalidomide base regimen in patients with relapsed or refractory DLBCL, with objective response rate as the primary end point.

DETAILED DESCRIPTION:
This study retrospectively collected the data of patients previously treated with Tafa and divided them into two coords according to different protocols received. Cohort 1 was Tafa combined treatment group, which could include Tafa combined with lenalidomide, Tafa combined with Lenalidomide plus BTK inhibitor, Tafa combined with Lenalidomide plus chemotherapy (including ADC). Cohort 2 was treated with sequential CAR T or graft after Tafa combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological diagnosis of DLBCL, including but not limited to non-specific DLBCL (NOS-DLBCL); Large B-cell lymphoma (THRLBCL) rich in T cells/histiocytes; EBV positive DLBCL (EBV-positive DLBCL); According to the revised REAL/WHO classification, it was grade 3b follicular lymphoma, including DLBCL component, followed by DLBCL recurrence. In addition, patients with low-grade lymphomas such as follicular lymphoma, marginal zone lymphoma, and chronic lymphocytic leukemia have histological evidence of transformation to DLBCL and subsequent recurrence
* Patients who, as determined by the treating physician, would benefit from Tafa treatment

Exclusion Criteria:

* Known allergy or metabolic disorder to any drug in the regimen
* Those who refuse to use reliable methods of contraception during pregnancy, lactation or age-appropriate period
* Have a history of uncontrolled medical disease (including uncontrolled diabetes, severe heart, lung, liver, renal insufficiency), blood, endocrine system, and other malignancies
* Severe mental illness
* Patients deemed unsuitable for inclusion by the investigator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recurrent or refractory diffuse large B-cell lymphoma after systemic therapy
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
objective remission rate | at the end of Cycle 2 (each cycle is 28 days)
  Defined as the proportion of patients with CR and PR

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1year after induction therapy
  The time between the start of treatment and when the tumor progresses or the patient dies

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided